CLINICAL TRIAL: NCT02584478
Title: A Phase 1/2a/3 Evaluation of the Safety and Efficacy of Adding AL3818 (Anlotinib, INN: Catequentinib), a Dual Receptor Tyrosine Kinase Inhibitor, to Standard Platinum-Based Chemotherapy in Subjects With Recurrent or Metastatic Endometrial, Ovarian, Fallopian, Primary Peritoneal or Cervical Carcinoma
Brief Title: Phase 1/2a/3 Evaluation of Adding AL3818 to Standard Platinum-Based Chemotherapy in Subjects With Recurrent or Metastatic Endometrial, Ovarian, Fallopian, Primary Peritoneal or Cervical Carcinoma (AL3818-US-002)
Acronym: AL3818
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Advenchen Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AL3818-US-002
Record Dates: First submitted 2015-08-28; First posted 2015-10-22 (Estimated); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Endometrial Carcinoma; Ovarian Carcinoma; Fallopian Tube Carcinoma; Primary Peritoneal Carcinoma; Cervical Carcinoma
Keywords: Dual receptor Tyrosine Kinase Inhibitor; Anti-angiogenic therapy; Combination Therapy
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms; Fallopian Tube Neoplasms; Uterine Cervical Neoplasms | interventions — anlotinib; Paclitaxel; liposomal doxorubicin; Topotecan; Carboplatin

STUDY DESIGN:
Intervention Model Description: Overall duration of the study will be approximately 42 months. Part 1 and 2 of this study are not randomized and have no concurrent controls. AL3818 and chemotherapy will be administered in an open-label fashion. Phase III/Part 3 is unblinded and randomized. Within each one of the three background chemotherapy groups, subjects will be randomized at a 1:1 ratio stratified by prior angiogenesis inhibitors mainly Avastin use status (Yes or No) and number of prior treatment (≤3 or >3) to receive AL3818 plus background chemotherapy (Active Arm) or background chemotherapy alone (Control Arm).
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase 3 -Active Treatment Arm (Experimental): Phase 3: AL3818 8 mg once daily in combination with one background chemotherapy in 21-day cycles. Platinum resistant recurrent or metastatic ovarian, fallopian, or primary peritoneal cancer subjects will be enrolled into one of the following three background chemotherapy groups:
  * Weekly paclitaxel (default choice; if the subject is ineligible for paclitaxel, the investigator will select from PLD or topotecan)
  * Pegylated liposomal doxorubicin (PLD)
  * Topotecan
  Interventions: Drug: AL3818; Drug: Paclitaxel; Drug: Pegylated Liposomal Doxorubicin (PLD); Drug: Topotecan
- Phase 3-Control Treatment Arm (Other): Control Treatment Arm: Background chemotherapy treatment alone. Platinum resistant recurrent or metastatic ovarian, fallopian, or primary peritoneal cancer subjects will be enrolled into one of the following three background chemotherapy groups:
  * Weekly paclitaxel (default choice; if the subject is ineligible for paclitaxel, the investigator will select from PLD or topotecan)
  * Pegylated liposomal doxorubicin (PLD)
  * Topotecan
  Interventions: Drug: Paclitaxel; Drug: Pegylated Liposomal Doxorubicin (PLD); Drug: Topotecan
- Phase 1b: AL3818 plus carboplatin and paclitaxel (Experimental): Phase 1b: Sequential deescalating dosing evaluation to determine the recommended Phase II dose (RP2D). For 21-day treatment cycles, cohort 1 (3 subjects) will be administered carboplatin (AUC 5/6 over 30 minutes) and paclitaxel (175mg/m2 over 3 hours) intravenously on Day 1. AL3818 is orally administered daily starting on Day 8 until Day 21 (14 days) at an initial dose of 12 mg/day.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: AL3818
- Phase 2a: AL3818 plus carboplatin and paclitaxel (Experimental): Phase 2a: subjects will receive chemotherapy and oral AL3818 for 6 cycles (18 weeks, 21-day cycles of treatment) followed by continuous maintenance treatment of oral AL3818 for up to 12 months. Subjects will be administered carboplatin (AUC 5/6 over 30 minutes) and paclitaxel (175mg/m2 over 3 hours) intravenously on Day 1. AL3818 is orally administered daily starting on Day 8 until Day 21 (14 days) at the RP2D found in Phase 1b.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: AL3818

INTERVENTIONS:
Drug: AL3818 — Taken daily from Day 8 to Day 21 (14 days),administered orally combination with one background chemotherapy in 21-day cycles.
  Other Names: Anlotinib Hydrochloride; Anlotinib; Catequentinib
  Arms: Phase 3 -Active Treatment Arm
Drug: Paclitaxel — Weekly single agent Paclitaxel will be administered on Day 1, 8, and 15 of each 21-day cycle. Suggested dose: 80 mg/m^2 intravenously or local standard.
  Paclitaxel may also be administered once weekly with a 1-week break every 3 weeks in lieu of every week
  Arms: Phase 3 -Active Treatment Arm; Phase 3-Control Treatment Arm
Drug: Pegylated Liposomal Doxorubicin (PLD) — Single agent Pegylated Liposomal Doxorubicin (PLD) administered every 4 weeks on the following cycle days corresponding with AL3818 cycles until maximum cumulative dose per local standard reached.
  Suggested dose: 40 mg/m^2 intravenously or local standard
  Arms: Phase 3 -Active Treatment Arm; Phase 3-Control Treatment Arm
Drug: Topotecan — Daily Topotecan on Days 1-5 of each 21-day cycle Suggested dose: 1.25 mg/m2 intravenously or local standard OR Weekly Topotecan with a 1 week break every 3 weeks. Suggested dose: 4 mg/m2 intravenously or local standard
  Other Names: Daily Topotecan
  Arms: Phase 3 -Active Treatment Arm; Phase 3-Control Treatment Arm
Drug: Topotecan — Weekly Topotecan with a 1 week break every 3 weeks Suggested dose: 4 mg/m2 intravenously or local standard
  Other Names: Weekly Topotecan
  Arms: Phase 3 -Active Treatment Arm; Phase 3-Control Treatment Arm
Drug: Carboplatin — AUC 5/6 on Day 1 of each 21-Day cycles
  Other Names: Paraplatin
  Arms: Phase 1b: AL3818 plus carboplatin and paclitaxel; Phase 2a: AL3818 plus carboplatin and paclitaxel
Drug: Paclitaxel — 175mg/m2 IV over 3 hours on Day 1 of each 21-Day cycle
  Other Names: Taxol
  Arms: Phase 1b: AL3818 plus carboplatin and paclitaxel; Phase 2a: AL3818 plus carboplatin and paclitaxel
Drug: AL3818 — Taken daily from Day 8 to Day 21 (14 days). Administered orally.
  Arms: Phase 1b: AL3818 plus carboplatin and paclitaxel; Phase 2a: AL3818 plus carboplatin and paclitaxel

SUMMARY:
This trial is a Phase 1b/2a/3 trial designed to evaluate the safety and efficacy of adding oral AL3818 (Anlotinib, INN: Catequentinib), a Dual Receptor Tyrosine Kinase Inhibitor, to standard platinum-based chemotherapy concurrently in Subjects with Recurrent or Metastatic Endometrial, Ovarian, Fallopian, Primary Peritoneal or Cervical Carcinoma.

DETAILED DESCRIPTION:
This trial is a Phase 1b/2a/3 trial designed to evaluate the safety and efficacy of adding oral AL3818(Anlotinib, INN: Catequentinib) to standard platinum-based chemotherapy concurrently and continued as a maintenance therapy for up to 12 months, in subjects with recurrent or metastatic endometrial, ovarian, fallopian, primary peritoneal, or cervical carcinoma. AL3818 is a novel small molecule dual receptor tyrosine kinase inhibitor, which shows highly selective inhibition of fibroblast growth factor receptor (FGFr) and vascular endothelial growth factor receptor (VEGFR). Preclinical studies of this agent in mouse models, including various cancer xenografts, have demonstrated that treatment of tumor-bearing mice with AL3818 induces tumor reductions.

Phase 1 & 2: This study is divided into two parts. The objective of Part 1 is the evaluation of the safety and tolerability of adding oral AL3818 to standard carboplatin plus paclitaxel chemotherapy for a cycle of 21 days to determine the recommended Phase II dose (RP2D). Phase 1 / Part 1 is now complete. Part 2-The objective of Part 2 is evaluation of preliminary efficacy and the safety of adding oral AL3818 at the RP2D determined in Part 1 to carboplatin and paclitaxel chemotherapy for 6 cycles. Continuous maintenance mono therapy with 14 days on and 7 days off regimen at the RP2D will be conducted up to 12 months and is extendable beyond until disease progression. Phase I is closed and Phase 2 is closed.

Phase 3: This study is currently a Phase III, multi-center, randomized trial with active control designed to evaluate the efficacy and safety of AL3818 8 mg plus background treatment (Active Arm) vs background treatment alone (Control Arm), where three background treatments, weekly paclitaxel, pegylated liposomal doxorubicin (PLD), and topotecan are utilized. Oral AL3818 8 mg may be given concurrently with background treatment or alone if the background treatment must be discontinued due to its toxicity for up to 24 cycles of therapy, in subjects with recurrent or metastatic platinum-resistant ovarian, fallopian tube, or primary peritoneal cancer. Phase 3 is open.

ELIGIBILITY:
Inclusion Critera

1. Female ≥ 18 years of age
2. Histologically proven diagnosis of:

   a. Endometrial and other uterine cancers with tumors of all histologies i. Recurrent Stage I to II endometrial and other uterine cancers, after at least one prior line of standard therapy, requiring further treatment with platinum-based chemotherapy ii. Advanced Stage III to IV endometrial and other uterine cancers requiring treatment with platinum-based chemotherapy

   b. Ovarian Cancer: Platinum-sensitive or platinum-resistant recurrent or metastatic ovarian, fallopian, or primary peritoneal cancer treated with at least one prior line of platinum-based chemotherapy and requiring further treatment.(Part 1/Phase Ib, Part 2/Phase 2a)

   Platinum-sensitive is defined as cancer progression ≥ 6 months after platinum- based chemotherapy. Platinum-resistant is defined as cancer progression < 6 months after platinum-based chemotherapy.

   Histologic cell types eligible are endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified.

   Phase III/Part 3:

(1) Platinum-resistant (progression within 6 months after last platinum-based chemotherapy) ovarian, fallopian, or primary peritoneal cancer that meets one of the following criteria: i. Subject has received at least two prior lines of systemic therapy including a bevacizumab-containing regimen as standard of care ii. Subject has received at least two prior lines of systemic therapy, has not received a prior bevacizumab-containing regimen and is not eligible for a bevacizumab containing regimen based on Investigator's assessment (2) Platinum-refractory (progression during first-line platinum-based chemotherapy) ovarian, fallopian, or primary peritoneal cancer after at least one prior line of systemic therapy (3) For groups 1-2 above: Subjects with positive deleterious or suspected deleterious, germline or somatic BRCA mutated status must have received a PARP inhibitor as a prior line of therapy.

c. Cervical cancer: recurrent or metastatic cervical cancer that is not amenable to curative treatment with surgery and/or radiation therapy after at least one prior line of standard therapy, requiring further treatment. Histologic cell types eligible are squamous cell carcinoma, adenosquamous carcinoma or adenocarcinoma

3. Have measureable disease defined by RECIST 1.1 confirmed by CT or MRI scan within 28 days of enrollment.

4. Life expectancy of ≥ 3 months at the time of enrollment.

5. Able to take orally administered study medication.

6. Have adequate baseline function and performance status within 28 days of enrollment:

1. Bone marrow function: absolute neutrophil count (ANC) ≥ 1,500/mm3, platelets ≥ 100,000/mm3
2. Renal function: creatinine ≤ 1.5 x institutional upper limit normal (ULN) or if creatinine is > 1.5 x ULN, creatinine clearance must be > 50 mL/min.
3. Hepatic function: bilirubin ≤ 1.5 x ULN or ≤ 3.0 x ULN for subjects with Gilbert Syndrome; AST and ALT ≤ 3.0 × ULN.
4. Coagulation profile: international normalized ratio (INR) is ≤ 1.5 and an aPTT or PTT < 1.2 x ULN
5. ECOG performance ≤ 2

   7. Women of child-bearing potential must agree to use contraceptive measures starting 1 week before C1D1 until 4 weeks after the last dose of study treatment and have a negative serum pregnancy test within 28 days of enrollment.

   8. Provide written informed consent and authorization permitting release of Protected Health Information.

   9. Ability and willingness to comply with the study protocol for the duration of the study and with follow-up procedures.

Exclusion Criteria

1. Serious, non-healing wound, ulcer or bone fracture.
2. Major surgical procedure within 28 days or minor surgical procedure performed within 7 days prior to C1D1 (a major surgical procedure is defined as requiring general anesthesia).
3. (Intentionally left blank)
4. Active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels.
5. History or evidence upon physical examination of central nervous system (CNS) disease including primary brain tumor; seizures not controlled with standard medical therapy; and history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA), or subarachnoid hemorrhage within 6 months of enrollment.

   a. Subjects with metastatic CNS tumors may participate in this study if the subject is > 28 days from therapy completion (including radiation and/or surgery), is clinically stable at the time of study enrollment, and is not receiving corticosteroid therapy.
6. Proteinuria on urinalysis within 28 days of enrollment. Subjects discovered to have a urine protein of 1+ on dipstick or ≥ 30 mg/dl at baseline should undergo a 24-hour urine collection and demonstrate < 1000 mg protein per 24 hours or spot urine protein (mg/dL) to creatinine (mg/dL) ratio must be <1.0 to allow participation in the study.
7. Clinically significant cardiovascular disease including uncontrolled hypertension; myocardial infarction or unstable angina within 6 months prior to enrollment; New York Heart Association (NYHA) Grade II or greater congestive heart failure (Appendix E); serious cardiac arrhythmia requiring medication; and Grade II or greater peripheral vascular disease.
8. Women who are pregnant or nursing.
9. (Intentionally left blank)
10. Clinically significant, uncontrolled hypokalemia, hypomagnesaemia, and/or hypocalcaemia.
11. Hemoptysis within 3 months prior to enrollment.
12. Acute or chronic liver disease, active hepatitis A or B with known cirrhosis or liver dysfunction.
13. Cytotoxic chemotherapy, immunotherapy, or radiotherapy within 28 days (42 days in cases of mitomycin C, nitrosourea, lomustine) prior to enrollment.
14. Concomitant treatment with strong inhibitors or inducers of CYP3A4, CYP2C9 and CYP2C19 within 14 days prior to enrollment and during the study unless there is an emergent or life-threatening medical condition that required it.
15. Known history of human immunodeficiency virus infection (HIV).
16. Active bacterial infections requiring systemic antibiotics (excluding uncomplicated urinary tract infection).
17. Other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of other cancer present within the last 5 years prior to enrollment or whose previous cancer treatment contraindicates this protocol therapy.
18. History of non-malignant gastrointestinal bleeding, gastric stress ulcerations, or peptic ulcer disease within the past 3-months prior to enrollment that in the opinion of the investigator may place the subject at risk of side effects on an anti-angiogenesis product.
19. History of significant vascular disease (e.g. aortic aneurysm, aortic dissection).
20. Intra-abdominal abscess within the last 3 months of enrollment.
21. Pre-existing uncontrolled hypertension as documented by two baseline blood pressure readings taken at least five minutes apart, defined as systolic BP >160 mm Hg or diastolic BP > 90 mm Hg pressure.
22. QTc > 470 msec on screening ECG per Fridericia's formula.
23. History of or existing risk factors for Torsades de pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
24. Concurrent use of concomitant medications that prolong the QT/QTc interval.
25. Baseline echocardiogram (within 56 days of enrollment) with left ventricular ejection fraction (LVEF) < 50%.
26. History of difficulty swallowing, malabsorption, active partial or complete bowel obstruction, or other chronic gastrointestinal disease or condition that may hamper compliance and/or absorption of AL3818.
27. History of pancreatitis; history of renal disease that includes histologically confirmed glomerulonephritis, biopsy proven tubulointerstitial nephritis, crystal nephropathy or other renal insufficiencies.
28. Treatment with an investigational agent within 28 days of enrollment.
29. Known recreational substance abuse.
30. Anticoagulation therapy with warfarin. Subjects treated with heparin, low molecular weight heparin, or any other anticoagulant may be included provided the subject has been on a stable therapeutic dose of the anticoagulant for at least 14 days prior to enrollment.
31. Known hypersensitivity to AL3818 or components of the formulation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2015-12; Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) - Part 1 (Phase 1b) | Cycle 1 (21-days)
  Determine the Recommended Phase 2 Dose (RP2D) via evaluation of dose limiting toxicity (DLT) events.
Objective Response Rates (ORR) - Part 2 (Phase 2a) | 12 months
  Evaluated by Response Evaluation Criteria In Solid Tumors (RECIST, v1.1) criteria after three complete 21-day cycles in the first 9 cycles then once every 6 cycles for up to 12 months. ORR is measured by the number of complete (CR) and partial responses (PR)
Measure the Progression Free Survival (PFS)- Part 3 ( Phase 3) | 12 Months
  To evaluate the efficacy between the Active Arm (AL3818 in combination with background chemotherapy) and Control Arm (background chemotherapy alone arm) as measured by the primary endpoint of Progression Free Survival (PFS).

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a measure of safety and toxicity of 21-Day cycles of AL3818 as measured by incidence and severity of treatment-related adverse events (TRAE) - Part 1 (Phase 1b) | Cycle 1 (Day 21)
  Incidence and severity of treatment-related adverse events reported and their relationship to AL3818 will be assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.3).
Clinical Benefit Rate (CBR) - Part 2 (Phase 2a) | 12 Months
  Evaluated by Response Evaluation Criteria In Solid Tumors (RECIST, v1.1) criteria after three complete 21-day cycles in the first 9 cycles then once every 6 cycles for up to 12 months. Measured as CR+PR+SD (SD ≥ 16 weeks from inclusion).
Progression-Free Survival (PFS) - Part 2 (Phase 2a) | Duration of time from the start of treatment to the time of documented disease progression or death, whichever comes first, followed for 12 months.
  Evaluated by Response Evaluation Criteria In Solid Tumors (RECIST, v1.1) criteria after three complete 21-day cycles in the first 9 cycles then once every 6 cycles for up to 12 months. Kaplan-Meier analysis
Overall Survival (OS) - Part 2 (Phase 2a) | Cycle 1 Day 1 up to 5 years
  Overall survival is defined as the date the study treatment was initiated to the date of death from any cause. Kaplan-Meier analysis
Objective Response Rate- Part 3 ( Phase 3) | 12 Months
  To evaluate the efficacy between the Active Arm and Control Arm as measured by the secondary endpoints of objective response rate (ORR). (OS).
Duration Of Response - Part 3 ( Phase 3) | 12 Months
  To evaluate the efficacy between the Active Arm and Control Arm as measured by the secondary endpoints of duration of response (DOR)
Overall Survival - Part 3 ( Phase 3) | 12 Months
  To evaluate the efficacy between the Active Arm and Control Arm as measured by the endpoints of Overall survival

OTHER OUTCOMES:
Toxicity as assessed by CTCAE (v4.3) - Part 2 (Phase 2a) | 12 Months
  Incidence and severity of treatment-related adverse events reported and their relationship to AL3818 will be assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.3)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, Study Director — Advenchen Laboratories, LLC
Locations (41):
- United States (8):
  - The Oncology Institute of Hope and Innovation, Long Beach, California
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Baptist Health Lexington Oncology Research, Lexington, Kentucky
  - Washington University, St Louis, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - AHN West Penn Hospital, Pittsburgh, Pennsylvania
  - UTSW, Dallas, Texas
  - University of Wisconsin Madison, Madison, Wisconsin
- China (9):
  - Henan Cancer Hospital, Hefei, Henan
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Shenyang
  - Zhongda Hospital Southeast University, Chongqing, Sichuan
  - Tianjin Central Hospital of Gynecology Obstetrics, Tianjin, Tianjin Municipality
  - Obstetrics&Gynecology Hospital of Fudan University, Shanghai, Yangpu District
  - Beijing Cancer Hospital, Beijing
  - Chongqing University Cancer Hospital, Chongqing
  - Weifang People's Hospital, Weifang
- Italy (8):
  - National Cancer Institute IRCCS "G. Pascale" Foundation, Naples, Campania
  - University Hospital of Bologna-IRCCS, Bologna, Emilia-Romagna
  - Romagnolo Institute For the Study of Tumors "Dino Amadori", Meldola (FC), Forlì-Cesena
  - Cannizzaro Emergency Hospital, Catania
  - Complex Structure Gynecology Oncology National Cancer Institute of Milan, Milan
  - Operative Unit of Oncology, Ravenna
  - Agostino Gemelli University Hospital Rome, Rome
  - Campus Bio Medico University Hospital Foundation, Rome
- South Korea (4):
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
- Spain (9):
  - Hospital Universitario Reina Sofía, Córdoba, Andalusia
  - Hospital Regional Universitario de Málaga, Málaga, Andalusia
  - ICO Badalona, Badalona, Catalonia
  - Hospital Universitari Vall d'Hebrón, Barcelona, Catalonia
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - HCU Virgen Arrixaca, Murcia
- United Kingdom (3):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Background] Hoeben A, Landuyt B, Highley MS, Wildiers H, Van Oosterom AT, De Bruijn EA. Vascular endothelial growth factor and angiogenesis. Pharmacol Rev. 2004 Dec;56(4):549-80. doi: 10.1124/pr.56.4.3. PMID 15602010
- [Background] Kondo Y, Arii S, Mori A, Furutani M, Chiba T, Imamura M. Enhancement of angiogenesis, tumor growth, and metastasis by transfection of vascular endothelial growth factor into LoVo human colon cancer cell line. Clin Cancer Res. 2000 Feb;6(2):622-30. PMID 10690548
- [Background] Roskoski R Jr. Vascular endothelial growth factor (VEGF) signaling in tumor progression. Crit Rev Oncol Hematol. 2007 Jun;62(3):179-213. doi: 10.1016/j.critrevonc.2007.01.006. Epub 2007 Feb 26. PMID 17324579
- [Background] Dickson C, Spencer-Dene B, Dillon C, Fantl V. Tyrosine kinase signalling in breast cancer: fibroblast growth factors and their receptors. Breast Cancer Res. 2000;2(3):191-6. doi: 10.1186/bcr53. Epub 2000 Mar 25. PMID 11250709
- [Background] Cole C, Lau S, Backen A, Clamp A, Rushton G, Dive C, Hodgkinson C, McVey R, Kitchener H, Jayson GC. Inhibition of FGFR2 and FGFR1 increases cisplatin sensitivity in ovarian cancer. Cancer Biol Ther. 2010 Sep 1;10(5):495-504. doi: 10.4161/cbt.10.5.12585. Epub 2010 Sep 4. PMID 20595807
- [Background] Raja FA, Griffin CL, Qian W, Hirte H, Parmar MK, Swart AM, Ledermann JA. Initial toxicity assessment of ICON6: a randomised trial of cediranib plus chemotherapy in platinum-sensitive relapsed ovarian cancer. Br J Cancer. 2011 Sep 27;105(7):884-9. doi: 10.1038/bjc.2011.334. Epub 2011 Aug 30. PMID 21878941
- [Background] Ledermann JA, Perren TJ, Raja FA, et al: Randomized double-blind phase III trial of cediranib (AZD 2171) in relapsed platinum-sensitive ovarian cancer: Results of the ICON6 trial. European Cancer Congress. Abstract 10. Presented September 30, 2013.
- [Background] Niu G, Chen X. Vascular endothelial growth factor as an anti-angiogenic target for cancer therapy. Curr Drug Targets. 2010 Aug;11(8):1000-17. doi: 10.2174/138945010791591395. PMID 20426765
- [Background] Shen GH, Ghazizadeh M, Kawanami O, Shimizu H, Jin E, Araki T, Sugisaki Y. Prognostic significance of vascular endothelial growth factor expression in human ovarian carcinoma. Br J Cancer. 2000 Jul;83(2):196-203. doi: 10.1054/bjoc.2000.1228. PMID 10901370
- [Background] Chen CA, Cheng WF, Lee CN, Chen TM, Kung CC, Hsieh FJ, Hsieh CY. Serum vascular endothelial growth factor in epithelial ovarian neoplasms: correlation with patient survival. Gynecol Oncol. 1999 Aug;74(2):235-40. doi: 10.1006/gyno.1999.5418. PMID 10419737
- [Background] Yoneda J, Kuniyasu H, Crispens MA, Price JE, Bucana CD, Fidler IJ. Expression of angiogenesis-related genes and progression of human ovarian carcinomas in nude mice. J Natl Cancer Inst. 1998 Mar 18;90(6):447-54. doi: 10.1093/jnci/90.6.447. PMID 9521169
- [Background] Cannistra SA, Matulonis UA, Penson RT, Hambleton J, Dupont J, Mackey H, Douglas J, Burger RA, Armstrong D, Wenham R, McGuire W. Phase II study of bevacizumab in patients with platinum-resistant ovarian cancer or peritoneal serous cancer. J Clin Oncol. 2007 Nov 20;25(33):5180-6. doi: 10.1200/JCO.2007.12.0782. PMID 18024865
- [Background] Burger RA, Brady MF, Bookman MA et al. Phase III trial of bevacizumab (BEV) in the primary treatment of advanced epithelial ovarian cancer (EOC), primary peritoneal cancer (PPC) or fallopian tube cancer (FTC): A Gynecologic Oncology Group study. Journal of Clinical Oncology, 2010 ASCO Annual Meeting Proceedings. Vol. 28, No 18S, 2010 June 20 suppl: Abstract LBA1
- [Background] Aghajanian C, Blank SV, Goff BA, Judson PL, Teneriello MG, Husain A, Sovak MA, Yi J, Nycum LR. OCEANS: a randomized, double-blind, placebo-controlled phase III trial of chemotherapy with or without bevacizumab in patients with platinum-sensitive recurrent epithelial ovarian, primary peritoneal, or fallopian tube cancer. J Clin Oncol. 2012 Jun 10;30(17):2039-45. doi: 10.1200/JCO.2012.42.0505. Epub 2012 Apr 23. PMID 22529265
- [Background] Yokoyama Y, Charnock-Jones DS, Licence D, Yanaihara A, Hastings JM, Holland CM, Emoto M, Sakamoto A, Sakamoto T, Maruyama H, Sato S, Mizunuma H, Smith SK. Expression of vascular endothelial growth factor (VEGF)-D and its receptor, VEGF receptor 3, as a prognostic factor in endometrial carcinoma. Clin Cancer Res. 2003 Apr;9(4):1361-9. PMID 12684405
- [Background] Holland CM, Day K, Evans A, Smith SK. Expression of the VEGF and angiopoietin genes in endometrial atypical hyperplasia and endometrial cancer. Br J Cancer. 2003 Sep 1;89(5):891-8. doi: 10.1038/sj.bjc.6601194. PMID 12942123
- [Background] Giatromanolaki A, Sivridis E, Brekken R, Thorpe PE, Anastasiadis P, Gatter KC, Harris AL, Koukourakis MI; Tumour and Angiogenesis Research Group. The angiogenic "vascular endothelial growth factor/flk-1(KDR) receptor" pathway in patients with endometrial carcinoma: prognostic and therapeutic implications. Cancer. 2001 Nov 15;92(10):2569-77. doi: 10.1002/1097-0142(20011115)92:103.0.co;2-3. PMID 11745191
- [Background] Gornall RJ, Anthony FW, Coombes EJ, Hogston P, Woolas RP. Investigation of women with endometrial carcinoma using serum vascular endothelial growth factor (VEGF) measurement. Int J Gynecol Cancer. 2001 Mar-Apr;11(2):164-6. doi: 10.1046/j.1525-1438.2001.011002164.x. PMID 11328416
- [Background] McMeekin DS, Sill MW, Benbrook D, Darcy KM, Stearns-Kurosawa DJ, Eaton L, Yamada SD; Gynecologic Oncology Group. A phase II trial of thalidomide in patients with refractory endometrial cancer and correlation with angiogenesis biomarkers: a Gynecologic Oncology Group study. Gynecol Oncol. 2007 May;105(2):508-16. doi: 10.1016/j.ygyno.2007.01.019. Epub 2007 Feb 15. PMID 17306350
- [Background] Talvensaari-Mattila A, Soini Y, Santala M. VEGF and its receptors (flt-1 and KDR/flk-1) as prognostic indicators in endometrial carcinoma. Tumour Biol. 2005 Mar-Apr;26(2):81-7. doi: 10.1159/000085589. Epub 2005 May 3. PMID 15867479
- [Background] Saito M, Sato Y, Watanabe J, Kuramoto H, Kaba S, Fukuda T. Angiogenic factors in normal endometrium and endometrial adenocarcinoma. Pathol Int. 2007 Mar;57(3):140-7. doi: 10.1111/j.1440-1827.2006.02071.x. PMID 17295646
- [Background] Hirai M, Nakagawara A, Oosaki T, Hayashi Y, Hirono M, Yoshihara T. Expression of vascular endothelial growth factors (VEGF-A/VEGF-1 and VEGF-C/VEGF-2) in postmenopausal uterine endometrial carcinoma. Gynecol Oncol. 2001 Feb;80(2):181-8. doi: 10.1006/gyno.2000.6056. PMID 11161857
- [Background] Giatromanolaki A, Koukourakis MI, Turley H, Sivridis E, Harris AL, Gatter KC; Tumour and Angiogenesis Research Group. Phosphorylated KDR expression in endometrial cancer cells relates to HIF1alpha/VEGF pathway and unfavourable prognosis. Mod Pathol. 2006 May;19(5):701-7. doi: 10.1038/modpathol.3800579. PMID 16557278
- [Background] Aghajanian C, Sill MW, Darcy KM, Greer B, McMeekin DS, Rose PG, Rotmensch J, Barnes MN, Hanjani P, Leslie KK. Phase II trial of bevacizumab in recurrent or persistent endometrial cancer: a Gynecologic Oncology Group study. J Clin Oncol. 2011 Jun 1;29(16):2259-65. doi: 10.1200/JCO.2010.32.6397. Epub 2011 May 2. PMID 21537039
- [Background] Guidi AJ, Abu-Jawdeh G, Berse B, Jackman RW, Tognazzi K, Dvorak HF, Brown LF. Vascular permeability factor (vascular endothelial growth factor) expression and angiogenesis in cervical neoplasia. J Natl Cancer Inst. 1995 Aug 16;87(16):1237-45. doi: 10.1093/jnci/87.16.1237. PMID 7563170
- [Background] Wiggins DL, Granai CO, Steinhoff MM, Calabresi P. Tumor angiogenesis as a prognostic factor in cervical carcinoma. Gynecol Oncol. 1995 Mar;56(3):353-6. doi: 10.1006/gyno.1995.1062. PMID 7535719
- [Background] Ravazoula P, Zolota V, Hatjicondi O, Sakellaropoulos G, Kourounis G, Maragoudakis ME. Assessment of angiogenesis in human cervical lesions. Anticancer Res. 1996 Nov-Dec;16(6B):3861-4. PMID 9042271
- [Background] Dellas A, Moch H, Schultheiss E, Feichter G, Almendral AC, Gudat F, Torhorst J. Angiogenesis in cervical neoplasia: microvessel quantitation in precancerous lesions and invasive carcinomas with clinicopathological correlations. Gynecol Oncol. 1997 Oct;67(1):27-33. doi: 10.1006/gyno.1997.4835. PMID 9345352
- [Background] Cella DF. Manual for the Functional Assessment of Cancer Therapy (FACT) Measurement System (version 4). Center for Outcomes, Research and Education (CORE), Northwestern University, Chicago, 1997
- [Background] Wright JD, Viviano D, Powell MA, Gibb RK, Mutch DG, Grigsby PW, Rader JS. Bevacizumab combination therapy in heavily pretreated, recurrent cervical cancer. Gynecol Oncol. 2006 Nov;103(2):489-93. doi: 10.1016/j.ygyno.2006.03.023. Epub 2006 May 2. PMID 16647106
- [Background] 36. Krishnansu Sujata Tewari, Michael Sill, Harry J. Long,et al. Plenary Session, Abstract # 3, J Clin Oncol 31, 2013 (suppl; abstract 3)
- [Background] Pectasides D, Xiros N, Papaxoinis G, Pectasides E, Sykiotis C, Koumarianou A, Psyrri A, Gaglia A, Kassanos D, Gouveris P, Panayiotidis J, Fountzilas G, Economopoulos T. Carboplatin and paclitaxel in advanced or metastatic endometrial cancer. Gynecol Oncol. 2008 May;109(2):250-4. doi: 10.1016/j.ygyno.2008.01.028. Epub 2008 Mar 4. PMID 18299146
- [Background] Tinker AV, Bhagat K, Swenerton KD, Hoskins PJ. Carboplatin and paclitaxel for advanced and recurrent cervical carcinoma: the British Columbia Cancer Agency experience. Gynecol Oncol. 2005 Jul;98(1):54-8. doi: 10.1016/j.ygyno.2005.03.037. PMID 15904950
- [Background] Parmar MK, Ledermann JA, Colombo N, du Bois A, Delaloye JF, Kristensen GB, Wheeler S, Swart AM, Qian W, Torri V, Floriani I, Jayson G, Lamont A, Trope C; ICON and AGO Collaborators. Paclitaxel plus platinum-based chemotherapy versus conventional platinum-based chemotherapy in women with relapsed ovarian cancer: the ICON4/AGO-OVAR-2.2 trial. Lancet. 2003 Jun 21;361(9375):2099-106. doi: 10.1016/s0140-6736(03)13718-x. PMID 12826431
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961